CLINICAL TRIAL: NCT02687906
Title: An Open Label, Dose-finding, Pharmacokinetics, Safety, and Tolerability Study of a Single Dose Infusion of VABOMERE (Meropenem-Vaborbactam) in Pediatric Subjects From Birth to Less Than 18 Years of Age With Serious Bacterial Infections
Brief Title: Dose-finding, Pharmacokinetics, and Safety of VABOMERE in Pediatric Subjects With Bacterial Infections
Acronym: TANGOKIDS
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rempex (a wholly owned subsidiary of Melinta Therapeutics, LLC) (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: Melinta Therapeutics, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Rempex 507; 2016-000656-99 (EudraCT Number)
Record Dates: First submitted 2016-02-17; First posted 2016-02-22 (Estimated); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — meropenem and vaborbactam; vaborbactam; Carbapenems; beta-Lactamase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single dose IV meropenem-vaborbactam (Experimental): Vabomere (meropenem-vaborbactam) for IV injection will be administered as a single dose diluted in normal saline infused IV over 3 hours
  * Cohort 1 (n=8): 12 to < 18 years of age (40 mg/kg)
  * Cohort 2 (n=8): 6 to < 12 years of age (40 mg/kg)
  * Cohort 2b (n=4): 6 to < 12 years of age (60 mg/kg)
  * Cohort 3 (n=8): 2 to < 6 years of age (60 mg/kg)
  * Cohort 4 (n=8): 3 months to < 2 years of age (60 mg/kg)
  * Cohort 5 (n=24): Birth to < 3 months of age (dose TBD)
    * Group A: Gestational Age (GA) < 32 weeks, Postnatal Age (PNA) < 2 weeks (n=6)
    * Group B: GA < 32 weeks, PNA > 2 weeks (n=6)
    * Group C: GA > 32 weeks, PNA < 2 weeks (n=6)
    * Group D: GA > 32 weeks, PNA > 2 weeks (n=6)
  * Cohort 6 (n=7): 2 to < 12 years of age and ≤ 35 kg of weight (80 mg/kg)
  Interventions: Drug: Vabomere

INTERVENTIONS:
Drug: Vabomere — Vabomere (meropenem-vaborbactam) for IV injection
  Other Names: Combination meropenem and vaborbactam; carbapenem and beta-lactamase inhibitor

SUMMARY:
A single dose infusion of Vabomere (meropenem-vaborbactam) is being tested for dose-finding, pharmacokinetics, safety, and tolerability in pediatric subjects from birth to less than 18 years of age with serious bacterial infections

DETAILED DESCRIPTION:
In the current era of increased resistance to extended spectrum cephalosporins, carbapenem antimicrobial agents are frequently the antibiotics of "last defense" for the most resistant pathogens in serious infections, including those found in complicated Urinary Tract Infections (cUTI). The recent dissemination of serine carbapenemases (e.g. KPC) in Enterobacteriaceae in many hospitals worldwide now poses a considerable threat to the carbapenems and other members of the beta-lactam class of antimicrobial agents.

Rempex developed meropenem-vaborbactam administered as a fixed combination by IV infusion, to treat serious Gram-negative infections, such as cUTIs, including those infections caused by bacteria resistant to currently available carbapenems.

This study is an open label, dose-finding, pharmacokinetics, safety, and tolerability study of a single dose infusion of meropenem-vaborbactam in pediatric subjects from birth to less than 18 years of age with suspected or confirmed bacterial infection receiving antibiotic therapy or subjects receiving peri-operative prophylactic use of antibiotics.

ELIGIBILITY:
Inclusion Criteria:

1. A signed and dated written informed consent from the parent or legal representative and a subject assent (according to local IRB requirements);
2. Male or female from birth to < 18 years of age;
3. Are hospitalized, in stable condition, and receiving systemic antibiotics for a known or suspected bacterial infection; or subjects receiving peri-operative prophylactic use of antibiotics;
4. The subject will be observed in the hospital for at least 6 hours after the study drug is administered;
5. If female and has reached menarche, or has reached Tanner Stage 3 breast development (even if not having reached menarche), the subject is practicing appropriate birth control or is sexually abstinent;
6. Sufficient intravascular access (peripheral or central) to receive study drug.

Subjects will be excluded from the study if any of the following exclusion criteria apply prior to randomization:

1. Signs of severe sepsis including:

   1. Shock or profound hypotension that is not responsive to fluid challenge;
   2. Hypothermia (core temperature < 35.6 ºC or 96.1 ºF);
   3. Disseminated intravascular coagulation as evidenced by prothrombin time or partial thromboplastin time ≥ 2X the ULN or platelets < 50% of the lower limit of normal;
2. Any surgical or medical condition which, in the opinion of the investigator, would put the subject at increased risk or is likely to interfere with study procedures or PK of the study drug;
3. Females who are of childbearing potential and unwilling to practice abstinence or use at least two methods of contraception (oral contraceptives, barrier methods, approved contraceptive implant) during the entire study period;
4. Female adolescent subjects who are pregnant or breastfeeding or have a positive serum β-hCG pregnancy test at screening and at pre-dose Day 1;
5. Males who are unwilling to practice abstinence or use an acceptable method of broth control during the entire study period (i.e. condom with spermicide);
6. Renal function at screening as estimated by creatinine clearance < 50 mL/min /1.73 m^2 as calculated using the updated Schwartz bedside formula: eGFR = k x (height in cm) ÷ serum creatinine

   * k = 0.33 in pre-term infants.
   * k = 0.45 in term infants to 1 year of age.
   * k = 0.55 in children and adolescent girls.
   * k = 0.70 in adolescent boys.
7. Treatment within 30 days prior to enrollment with valproic acid;
8. Treatment within 30 days prior to enrollment with probenecid;
9. Evidence of significant hepatic disease or dysfunction, including known acute viral hepatitis or hepatic encephalopathy;
10. Neutropenia with absolute neutrophil count (ANC) < 500 cells/mm3;
11. Aspartate aminotransferase or alanine aminotransferase ≥ 3X ULN or total bilirubin ≥ 1.5X ULN;
12. Receipt of any investigational medication or investigational device within 30 days prior to enrollment;
13. Prior exposure to vaborbactam or Vabomere;
14. Use of meropenem within 48 hours of administration of study drug or 12 hours after study drug administration;
15. Known significant hypersensitivity to any beta-lactam antibiotic;
16. Unable or unwilling in the judgment of the Investigator, to comply with the protocol;
17. Subject is a child of an employee of the Investigator or study center with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as a family member of the employee or the Investigator;
18. Body Mass Index (BMI) outside the range (below the 5th percentile or above the 95th percentile) for height, age and weight except for children < 2 years of age.)

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics: AUC0-∞ | From pre-dose until 6 hours after the start of the infusion
  AUC from time zero to infinity
Pharmacokinetics: Cmax | From pre-dose until 6 hours after the start of the infusion
  maximum measured plasma concentration
Pharmacokinetics: time to maximum plasma concentration (Tmax) | From pre-dose until 6 hours after the start of the infusion
  time to Cmax
Pharmacokinetics: drug clearance (CL) | From pre-dose until 6 hours after the start of the infusion
  total body clearance
Pharmacokinetics: t1/2 | From pre-dose until 6 hours after the start of the infusion
  elimination half- life
Pharmacokinetics: Cmin | From pre-dose until 6 hours after the start of the infusion
  minimum plasma concentration
Pharmacokinetics: Vss | From pre-dose until 6 hours after the start of the infusion
  Volume of distribution
Safety and tolerability: AEs/SAEs | From assent / consent until day 7 safety follow up call
  a composite measure of the number and types of AEs/SAEs encountered and relationship to time of dosing
Safety and tolerability: clinical safety laboratory results | From assent / consent until day 7 safety follow up call
  A composite measure of multiple laboratory results assessing the clinical significance of any changes from baseline
Safety and tolerability: vital signs | From assent / consent until day 7 safety follow up call
  A composite of multiple vital sign measurements, assessing the clinical significance of any changes from baseline
Safety and tolerability: ECGs | From assent / consent until day 7 safety follow up call
  A composite of multiple ECG measurements, assessing the clinical significance of any changes from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Melinta Therapeutics, Inc.
Locations (9):
- United States (9):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Rutger's University, New Brunswick, New Jersey
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Toledo Children's Hospital, Toledo, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bradley JS, Harvey H, Stout D, Momper J, Capparelli E, Avedissian SN, Barbato C, Mak RH, Jones TP, Jones D, Le J. Subtherapeutic Meropenem Antibiotic Exposure in Children With Septic Shock Assessed by Noncompartmental Pharmacokinetic Analysis in a Prospective Dataset. Pediatr Crit Care Med. 2025 Apr 1;26(4):e507-e515. doi: 10.1097/PCC.0000000000003698. Epub 2025 Feb 18. PMID 39964222